CLINICAL TRIAL: NCT07363538
Title: Multicenter Randomized Controlled Trial (RCT) and Efficacy Evaluation System Study on Surgical Innovation Strategies for Neonatal Complex Congenital Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central China Fuwai Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Qihang Yang, postgraduate student, Central China Fuwai Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZD0527003
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Complex Congenital Heart Disease
MeSH Terms: interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Surgical operation is performed on neonates aged >7 days (postnatal age)
  Interventions: Procedure: Surgical operation is performed on neonates aged >7 days (postnatal age)
- Experimental Group (Experimental): Surgical operation is performed on neonates aged < 7 days (postnatal age)
  Interventions: Procedure: Surgical operation is performed on neonates aged < 7 days (postnatal age).

INTERVENTIONS:
Procedure: Surgical operation is performed on neonates aged >7 days (postnatal age) — Surgical operation is performed on neonates aged >7 days (postnatal age)
  Arms: Control Group
Procedure: Surgical operation is performed on neonates aged < 7 days (postnatal age). — Surgical operation is performed on neonates aged < 7 days (postnatal age).
  Arms: Experimental Group

SUMMARY:
There remains controversy regarding the optimal timing of surgical treatment for neonatal CCHD (Complex Congenital Heart Disease). Based on the established national multi-center database for surgical treatment of congenital heart disease and the prenatal-postnatal integrated diagnosis and treatment model, this study will conduct a multi-center RCT (Randomized Controlled Trial) to explore the optimal surgical timing for neonatal CCHD. It will also develop innovative comprehensive treatment strategies for critically ill neonatal CCHD patients, use RCT data to evaluate treatment efficacy and establish an evaluation system. This system will be gradually promoted nationwide, aiming to reduce the incidence of perioperative mortality and non-recovery discharge in CCHD patients by 50% (National in-hospital mortality rate of neonatal congenital heart disease surgery in 2023: 6.5%; non-recovery discharge rate: 12.66%), thereby improving the overall level of CCHD treatment in China.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates diagnosed with TAPVC, CoA/IAA, TGA, PA/IVS, or severe PS via pre-admission cardiac echocardiography;
2. Patients and families demonstrating high compliance, willing to sign informed consent forms and agree to complete one year of follow-up and related examinations.

Exclusion Criteria:

1. Preterm infant (gestational age < 36 weeks at birth);
2. Low birth weight (weight < 2.5 kg);
3. Concurrent severe extracardiac anomalies or complex cardiac malformations;
4. Preoperative respiratory or circulatory instability requiring emergency surgery.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 738 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative Mortality and Non-Rehabilitation Discharge Rate | From enrollment to 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou Medical University, Guangzhou, Guangdong
  - Central China Fuwai Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Children's Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Qingdao Women and Children's Hospital, Qingdao, Shandong
  - Shanghai Children's Medical Center (SCMC) Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Air Force Medical University (Xijing Hospital), Xi’an, Shanxi
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang